CLINICAL TRIAL: NCT06260033
Title: A Phase II Trial of Stereotactic Body Radiation Therapy and Fluoroestradiol Positron Emission Tomography in Patients With Oligoprogressive Estrogen Receptor Positive Metastatic Breast Cancer
Brief Title: Stereotactic Body Radiation Therapy and FES PET/CT Imaging for the Treatment of Oligoprogressive Estrogen Receptor Positive Metastatic Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23353; NCI-2023-11094 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23353 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2024-01-11; First posted 2024-02-15 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Estrogen Receptor-Positive Breast Carcinoma; Metastatic Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Specimen Handling; 16-fluoroestradiol; Magnetic Resonance Spectroscopy; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (SBRT, FES PET/CT) (Experimental): Patients currently taking SERMs/ SERDs immediately undergo 3 or 5 treatment fractions of SBRT within 3 weeks in the absence of unacceptable toxicity or evidence of > 4 sites of disease progression. Patients not currently taking SERMs/SERDs first receive F-FES IV and undergo PET/CT scans at baseline. After baseline FES PET/CT, patients with ≤ 4 sites of progressive disease then undergo 3 or 5 treatment fractions of SBRT within 3 weeks in the absence of unacceptable toxicity or evidence of > 4 sites of disease progression. All patients undergo FES PET/CT at 12 and 24 weeks. Patients with SD after 12 or 24 week FES PET/CT may continue standard systemic therapy. Patients with ≤ 4 sites of progressive disease after 12 or 24 week FES PET/CT may receive SBRT to additional sites in the absence of unacceptable toxicity or evidence of > 4 sites of disease progression. All patients also undergo CT, PET/CT, or bone scans, and blood samples collection during screening and on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Drug: F-18 16 Alpha-Fluoroestradiol; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
Procedure: Computed Tomography — Undergo PET/CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Drug: F-18 16 Alpha-Fluoroestradiol — Given IV
  Other Names: 16 alpha-fluroestradiol-17 beta; F-18 FES; FES; Fluorine-18 16 alpha-fluoroestradiol; Fluoroestradiol F-18
Procedure: Positron Emission Tomography — Undergo PET/CT scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Other: Questionnaire Administration — Ancillary studies
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy

SUMMARY:
This phase II trial tests how well stereotactic body radiation therapy (SBRT) works in treating patients with estrogen receptor positive (ER +) breast cancer that has spread from where it first started to other places in the body (metastatic) and has limited disease progression (oligoprogression). Currently, the standard of care for breast cancer patients with oligoprogressive disease is to change systemic therapy when progression occurs. Radiation therapy uses high energy x-rays, particles, or radioactive seeds to kill cancer cells and shrink tumors. SBRT is a type of external radiation therapy that uses special equipment to position a patient and precisely deliver radiation to tumors in the body (except the brain). The total dose of radiation is divided into smaller doses (fractions) given over several days. This type of radiation therapy helps spare normal tissue and has been shown to improve survival. SBRT may kill more tumor cells and allow patients with oligoprogressive ER + metastatic breast cancer to continue taking current systemic treatment.

This trial also tests how well ER targeted positron emission tomography (PET)/ computed tomography (CT) imaging, using FES, works in identifying progressive disease in patients with ER + metastatic breast cancer. FES, a radiolabeled substance, binds to estrogen receptors and gives off radiation that can be detected by a PET scan. The PET scan, an established imaging technique that utilizes small amounts of radioactivity attached to very minimal amounts of tracer, FES, forms an image that shows where tumor cells with estrogen receptors can be found in the body. CT images use x-rays to provide an exact outline of organs. FES PET/CT may improve identification of progressive disease in patients with ER + metastatic breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether using SBRT to treat oligoprogressive lesions allows ER+ breast cancer patients to continue on their current systemic therapy for at least 24 weeks post SBRT treatment.

SECONDARY OBJECTIVES:

I. To evaluate adverse events (Common Terminology Criteria in Adverse Events [CTCAE] and Patient-Reported Outcomes PRO-CTCAE) in patients who receive SBRT.

II. To assess whether F-18 16 alpha-fluoroestradiol (FES)-PET increases the number of lesions found prior to SBRT.

III. To determine the impact of SBRT on patient quality of life using the European Organization for the Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-C30 and QLQ-BR45.

IV. To estimate time to the next line of systemic therapy in patients who receive SBRT for oligoprogression.

V. To estimate progression-free survival time in patients who receive SBRT for oligoprogression.

EXPLORATORY OBJECTIVES:

I. To assess whether FES-PET increases the number of lesions found after SBRT. II. To describe circulating tumor deoxyribonucleic acid (ctDNA) levels over time after SBRT treatment.

III. To identify potential predictors of outcomes to treatment with SBRT.

OUTLINE:

Patients currently taking selective estrogen receptor modulators (SERMs)/selective estrogen receptor degraders (SERDs) immediately undergo 3 or 5 treatment fractions of SBRT within 3 weeks in the absence of unacceptable toxicity or evidence of > 4 sites of disease progression. Patients not currently taking SERMs/SERDs first receive F-FES intravenously (IV) and undergo PET/CT scans at baseline. After baseline FES PET/CT, patients with ≤ 4 sites of progressive disease then undergo 3 or 5 treatment fractions of SBRT within 3 weeks in the absence of unacceptable toxicity or evidence of > 4 sites of disease progression. All patients undergo FES PET/CT at 12 and 24 weeks. Patients with stable disease (SD) after 12 or 24 week FES PET/CT may continue standard systemic therapy. Patients with ≤ 4 sites of progressive disease after 12 or 24 week FES PET/CT may receive SBRT to additional sites in the absence of unacceptable toxicity or evidence of > 4 sites of disease progression. All patients also undergo CT, PET/CT, or bone scans, and blood samples collection during screening and on study.

After completion of study intervention, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative
* Age: ≥ 18 years
* Female or male
* Eastern Cooperative Oncology Group (ECOG) ≤ 2
* Ability to read and understand English or Spanish for questionnaires
* Histologically confirmed ER+ (any progesterone receptor [PR] and human epidermal growth factor receptor 2 [HER2] status is allowed) metastatic breast cancer
* The presence of metastatic breast cancer at the time of study entry with progression in 1-4 lesions (including new lesions). Patients that have disease progression in the breast and/or ipsilateral axilla will be considered to have only 1 site of progression even if multiple nodules/lymph nodes are present. Patients with progression in > 4 lesions are not allowed. Patients with current progression of malignant pleural effusions, malignant ascites, abdominal carcinomatosis, and/or lymphangitic pulmonary involvement are considered to have > 4 metastases (Note that patients with a history of these conditions earlier in the disease course with no evidence of progression of these conditions are eligible.)
* Evidence of extracranial disease progression in 1-4 discrete lesions will be defined by either of the following:

  * Progression of disease by Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1 or PET Response Criteria in Solid Tumors (PERCIST) v 1.0 criteria OR
  * Progression of disease in at least 1 but up to 4 lesions as determined by the patient's treating oncologists such that the treating oncologist recommends changing to the next line systemic therapy. Note that a patient may not technically meet RECIST v 1.1 criteria for disease progression in this setting
* SBRT must be feasible for all progressing lesions. Feasibility includes but is not limited to:

  * All progressing lesions must have distinct borders AND
  * Progressing lesions may not be located within 3 cm of previously irradiated critical structures such as the spinal cord, brachial plexus, brainstem, stomach, and/or small/large bowel that would render the metastasis unsafe to target with SBRT per the treating radiation oncologist
* Patients with prior treated brain metastases that are stable are allowed. Patients must not have intracranial disease progression. Patients with prior or current leptomeningeal disease are not allowed
* All progressing lesions must be amenable to stereotactic body radiation therapy to a dose of 30 Gy to 40 Gy in 3 to 5 fractions per the treating radiation oncologist
* Women of childbearing potential (WOCBP): Negative urine or serum pregnancy test, If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 1 months after the last dose of protocol therapy.

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* Has received at least one line, but not more than three lines, of systemic therapy for metastatic disease
* Patients may not have received chemotherapy, radiation therapy, biological therapy, immunotherapy, or other anti-cancer treatment within 7-14 days of the start of study therapy (SBRT) at the discretion of treating physician. Chemotherapy must be held during study therapy and can resume 7-14 days after completion of all study therapy (SBRT) at the discretion of treating physician. (Patients may continue anti-endocrine/hormone therapy before, during and after study therapy at the discretion of the treating medical oncologist.)
* Clinically significant uncontrolled illness such that the patient is no longer a candidate for systemic therapy
* Prior or concurrent malignancy. Prior malignancies with a low probability of recurrence requiring treatment such as the following are allowed: carcinoma in situ of the cervix, non-melanoma skin cancer, and low grade (Gleason score ≤ 6 = Gleason group 1) localized prostate cancer. Prior malignancies not listed require principal investigator (PI) approval
* Patients that have only liver metastases will not be allowed
* Females only: Pregnant or breastfeeding
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-07-23 (Actual); Primary Completion 2026-10-29 (Estimated); Study Completion 2026-10-29 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients that remain on their original systemic therapy for at least ≥ 24 weeks post stereotactic body radiation therapy (SBRT) treatment | Up to 24 weeks post SBRT treatment
  Analysis will be descriptive in nature and will include the counts and percentages of patients who are responders versus (vs.) non-responders. Results will summarize groups based on intent-to treat.

SECONDARY OUTCOMES:
Rate of all grades and grade ≥ 3 toxicities at least possibly related to study therapy | At baseline and post SBRT treatment up to 24 weeks
  Will be assessed by Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0 and patient reported outcomes CTCAE. Descriptive statistics will be used to summarize patient and physician reported toxicity. Results will be presented by entire group and stratified by response status (responders vs. non-responders). Chi-square analyses will be used to compare responders with non-responders at each timepoint.
Number of lesions found on F-18 16 alpha fluoroestradiol positron emission tomography (FES-PET) | At baseline prior to SBRT
  The number of additional lesions found on FES-PET prior to SBRT will be summarized using means, median, and ranges.
Change in quality of life (QOL) | At baseline and post SBRT treatment up to 24 weeks
  Descriptive statistics will be used to summarize changes in QOL measured using the European Organization for research and Treatment of Cancer Quality of Life Questionnaire Core 30 and Quality of Life Questionnaire Breast 45. Change from baseline results will be presented for the entire group as well as stratified by response status (responders vs. non-responders). Continuous data will be summarized using means and standard deviations, while categorical data will be summarized using counts and percentages. Difference across response status will be assessed using paired t-tests for continuous data and chi-square analyses for categorical data.
Time to next line of systemic therapy | At time from study entry up to next line of systemic therapy up to 24 weeks
  The time from next line of systemic therapy summarized using means, medians, and ranges and will be based on intent-to-treat. Time to next line of systemic therapy will be calculated from the date of study entry to the first date of next line therapy using the Kaplan-Meier method.
Progression free survival (PFS) | At time from study entry up to first occurrence of disease progression up to 24 weeks
  PFS will be assessed using Response Evaluation Criteria in Solid Tumors v 1.1 or Positron Emission Tomography Response Evaluation Criteria in Solid Tumors v 1.0. PFS will be summarized using means, medians, and ranges and will be based on intent-to-treat. PFS will be calculated from the date of study entry to the first date that progression was measured using the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Jose G Bazan, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - City of Hope at Irvine Lennar, Irvine, California